CLINICAL TRIAL: NCT03370510
Title: Translating Neuroprediction Into Precision Medicine Via Brain Priming
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Covid-19 Pandemic
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000021581
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Results first posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Eighty children will be randomly assigned to receive PRT with either oxytocin (forty children) or a placebo (forty children).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pivotal Response Treatment (PRT)/oxytocin (OXT) nasal spray (Experimental): Participants will receive oxytocin nasal spray 45 minutes prior to each PRT session.
  Interventions: Drug: Oxytocin; Behavioral: Pivotal Response Treatment
- Pivotal Response Treatment (PRT)/placebo nasal spray (Placebo Comparator): Participants will receive a placebo nasal spray 45 minutes prior to each PRT session.
  Interventions: Behavioral: Pivotal Response Treatment; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Oxytocin nasal spray.
  Arms: Pivotal Response Treatment (PRT)/oxytocin (OXT) nasal spray
Behavioral: Pivotal Response Treatment — An evidence-based manualized treatment for individuals with autism, which was specifically designed to improve social communication.
Drug: Placebo — Placebo nasal spray.
  Arms: Pivotal Response Treatment (PRT)/placebo nasal spray

SUMMARY:
The present study examines the impact of oxytocin (OXT) and Pivotal Response Treatment (PRT) on the development of language, social, and play skills in young children with Autism Spectrum Disorder (ASD). The purpose of this study is to examine the impact of OXT as an enhancer of response to PRT. Participants will be randomly assigned to either an intranasal OXT group or a placebo group. Neither the research team nor the participants will know or choose which group the participant is assigned to. Children in both groups will participate in a 16-week trial of PRT. The trial will test the hypothesis that children with lower levels of activity in and functional connectivity among certain PRT-response brain regions will benefit more from the administration of OXT vs. placebo as an enhancer to a 16-week trial of PRT.

DETAILED DESCRIPTION:
This project investigates the effectiveness of a new intervention approach for Autism Spectrum Disorder (ASD) to optimize the effects of an evidence-based behavioral intervention, Pivotal Response Treatment (PRT) by attempting to enhance it with oxytocin (OXT). We will integrate fMRI, eye tracking, and behavioral outcomes to measure how OXT may create a neural background for individuals with ASD to bolster their motivation to interact socially and facilitate their biological preparedness for learning social communication skills during behavioral treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Fit the age requirement: age 5-9
2. Have been diagnosed previously with an ASD and meet criteria for ASD when characterized by research team
3. Be in good medical health
4. Be cooperative with testing
5. Speak English in the family
6. Successfully complete an fMRI scan
7. Full-scale intelligence quotient (IQ)>70

Exclusion Criteria:

1. Any metal or electromagnetic implants, including:

   1. Cardiac pacemaker
   2. Defibrillator
   3. Artificial heart valve
   4. Aneurysm clip
   5. Cochlear implants
   6. Shrapnel
   7. Neurostimulators
   8. History of metal fragments in eyes or skin
2. Significant hearing loss or other severe sensory impairment
3. A fragile health status.
4. Current use of prescription psychotropic medications that may affect cognitive processes under study.
5. A history of significant head trauma or serious brain or psychiatric illness

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Sukhodolsky, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
Started | 3 | 2
Completed | 1 | 2
Not Completed | 2 | 0
Not completed — COVID-19 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Full Range); unit: Months] | 71 [62 to 89] | 82 [75 to 89] | 76 [62 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Social Responsiveness Scale, 2nd Edition (SRS-2)
Description: The SRS-2 is a 65-item measure of social responsiveness. The SRS-2 is filled out by a parent. The SRS-2 has a minimum raw score of 0 and a maximum raw score of 195. Higher raw scores on the SRS-2 mean a worse outcome.
Time Frame: Change from Baseline to post-treatment, 16 weeks
Population: Only 1/3 participants completed treatment in the oxytocin group. Therefore, the mean raw score for the oxytocin group is based off of that subject's data only.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
Number analyzed (Participants) | 1 | 2
score on a scale | 39 [39 to 39] | -16 [-21 to -11]

2. Secondary Outcome: Vineland Adaptive Behavior Scale, 3rd Edition (Vineland-III)
Description: The Vineland-III is a parent interview administered by a member of the research team. The interview lasts approximately one hour and measures four domains of the child's adaptive behavior.
Time Frame: Change from Baseline to post-treatment, 16 weeks
Population: Data were not collected due to COVID-19 related termination of study.
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Gaze Patterns
Description: Gaze patterns will be tracked using eye tracking technology as participants watch videos for approximately one hour.
Time Frame: Change from Baseline to post-treatment, 16 weeks
Population: Data were not collected due to COVID-19 related termination of study.
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Autism Diagnostic Observation Schedule - 2nd Edition (ADOS-2)
Description: The ADOS-2 is a diagnostic assessment for ASD performed by a clinician.
Time Frame: Change from Baseline to post-treatment, 16 weeks
Population: Data were not collected due to COVID-19 related termination of study.
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Clinical Global Impressions - Severity (CGI-S)
Description: The CGI-S is a 7-point Likert Scale completed by a clinician, which measures clinical impressions of symptom severity.
Time Frame: Change from Baseline to post-treatment, 16 weeks
Population: Data were not collected due to COVID-19 related termination of study.
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Social Responsiveness Scale - 2 (Teacher Form)
Description: The SRS-2 is a 65-item measure of social responsiveness. The SRS-2 Teacher is filled out by the participant's teacher.
Time Frame: Change from Baseline to post-treatment, 16 weeks
Population: Data were not collected due to COVID-19 related termination of study.
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Child Behavior Checklist (CBCL)
Description: The CBCL is a parent report measure of problem behaviors. The form for children ages 1.5-5 has 100 items, and the form for children ages 6-18 has 113 items.
Time Frame: Change from Baseline to post-treatment, 16 weeks
Population: Data were not collected due to COVID-19 related termination of study.
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Child and Adolescent Symptom Inventory - 5 (CASI-5)
Description: The CASI-5 is a behavior inventory measuring symptoms of several mental health problems among children. The CASI-5 is a 173-item parent report measure.
Time Frame: Change from Baseline to post-treatment, 16 weeks
Population: Data were not collected due to COVID-19 related termination of study.
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Aberrant Behavior Checklist (ABC)
Description: The ABC is a 58-item parent report behavior rating scale.
Time Frame: Change from Baseline to post-treatment, 16 weeks
Population: Data were not collected due to COVID-19 related termination of study.
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Repetitive Behavior Scale - Revised (RBS-R)
Description: The RBS-R is a 49-item, parent report measure of restricted and repetitive behaviors.
Time Frame: Change from Baseline to post-treatment, 16 weeks
Population: Data were not collected due to COVID-19 related termination of study.
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Behavior Rating Inventory of Executive Function (BRIEF)
Description: The BRIEF is an 86-item parent report measure of executive function.
Time Frame: Change from Baseline to post-treatment, 16 weeks
Population: Data were not collected due to COVID-19 related termination of study.
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Neural Activity/Connectivity During Videos of Biological Motion
Description: Neural activity while viewing videos of biological motion will be measured using fMRI.
Time Frame: Change from Baseline to post-treatment, 16 weeks
Population: Data were not collected due to COVID-19 related termination of study.
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Brief Observation of Social Communication Change (BOSCC)
Description: The BOSCC is a coding scheme that measures social communication change. Codes are based on videos of play session between children and parents.
Time Frame: Change from Baseline to post-treatment, 16 weeks
Population: Data were not collected due to COVID-19 related termination of study.
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Pivotal Response Treatment (PRT)/Oxytocin (OXT) Nasal Spray | Pivotal Response Treatment (PRT)/Placebo Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

LIMITATIONS AND CAVEATS:
This study was terminated early due to issues related to the covid-19 pandemic. Only 3 participants completed the trial- 1 out of 3 in the oxytocin group and 2 in the placebo group. As such, the mean score for the oxytocin group is based off of one subjects data only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT03370510/Prot_SAP_000.pdf